CLINICAL TRIAL: NCT00497588
Title: the Comparison of Voice Quality in Early Laryngeal Cancer Between Surgery and Radiotherapy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Babak Saedi, associate Professor, Tehran University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: bs-86-01-48-5497
Record Dates: First submitted 2007-07-04; First posted 2007-07-06 (Estimated); Last update posted 2013-07-11 (Estimated); Status verified 2013-07

CONDITIONS: Voice Quality
Keywords: laryngeal cancer; RADIOTHERAPY; Voice Quality
MeSH Terms: conditions — Laryngeal Neoplasms | interventions — Surgical Procedures, Operative; Radiotherapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- radiotherapy (Active Comparator): patients receive radiotherapy
  Interventions: Radiation: radiotherapy
- surgery (Experimental): Patients undergo surgery
  Interventions: Procedure: surgery

INTERVENTIONS:
Procedure: surgery
  Arms: surgery
Radiation: radiotherapy
  Arms: radiotherapy

SUMMARY:
early laryngeal cancer is a well known field with great controversy in treatment. two options are available in treatment of patients the first one is partial laryngectomy and the second one is radiotherapy.one of major concern of patients have been the quality of voice ,so we design this trial to answer the priority of each options.

DETAILED DESCRIPTION:
early laryngeal cancer is a well known field with great controversy in treatment. two options are available in treatment of patients the first one is partial laryngectomy and the second one is radiotherapy.one of major concern of patients have been the quality of voice as part of quality of life ,so we design this clinical randomised trial to answer the priority of each options.

ELIGIBILITY:
Inclusion Criteria:

* Early laryngeal cancer

Exclusion Criteria:

* No history of radiotherapy and collagen vascular disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2007-03; Primary Completion 2014-04 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
quality of voice | 3 to 6 month after therapy

SECONDARY OUTCOMES:
quality of life | 6 month later

CONTACTS AND LOCATIONS:
Overall Officials: babak saedi, professor, Principal Investigator — tehran university of medical science
Locations (1):
- Imam Khomainee hospital, Tehran, Tehran Province, Iran